CLINICAL TRIAL: NCT01488617
Title: Mainz Outcome Predictor Studies: An Observational Clinical Trial Investigating Physiological and Psychological Data as Predictors for Postoperative Outcome.
Brief Title: Mainz Outcome Predictor Studies: An Observational Clinical Trial Investigating Predictors for Postoperative Outcome
Acronym: MOPS
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Rita Laufenberg-Feldmann, M.D., Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: MOPS 2012
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Surgery; Psychological Distress
Keywords: Surgery; Psychosocial Factors; Psychological Distress; Outcome Assessment (Health Care)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether psychological and social factors in addition to medical (physiological) conditions may contribute significantly to the prediction of the postoperative outcome.

Postoperative outcome is defined (1) as postoperative complications and organ dysfunction and (2) alteration of quality of life.

DETAILED DESCRIPTION:
Different factors contribute to the recovery process after surgical intervention. However, little is known about the predictive value of single factors.

In addition to medical (physical) factors, depression, anxiety, somatization and avoiding coping styles are considered as relevant for the successful recovery process. These factors may be defined as "psychological distress" and could be used as predictors for perioperative complications and failed surgical treatment.

Postoperative outcome is defined (1) as postoperative complications and organ dysfunction and (2) alteration of quality of life.

Our sample includes adults undergoing extensive surgical interventions in trauma and orthopaedic surgery, urology, general surgery, and neurosurgery. The defined variables are measured using standardized and validated questionnaires prior to surgery and in follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Minimum Age 18 Years
* German language in speaking and writing
* Capability of giving consent
* written informed consent

Exclusion Criteria:

* Delirium, dementia or other mental disorders with significant cerebral dysfunction
* People under guardianship
* simultaneous participation in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients sceduled for elective surgery.
Sampling Method: Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | 6 weeks and 6 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Rita Laufenberg-Feldmann, M.D., Principal Investigator — Department of Anaesthesiology, University Medical Center of Johannes Gutenberg-University Mainz, Germany
Locations (1):
- Department of Anaesthesiology, University Medical Center of Johannes Gutenberg-University Mainz, Germany, Mainz, Germany

REFERENCES:
- [Derived] Laufenberg-Feldmann R, Kappis B, Camara RJA, Ferner M. Anxiety and its predictive value for pain and regular analgesic intake after lumbar disc surgery - a prospective observational longitudinal study. BMC Psychiatry. 2018 Mar 27;18(1):82. doi: 10.1186/s12888-018-1652-8. PMID 29587759
- [Derived] Laufenberg-Feldmann R, Kappis B, Mauff S, Schmidtmann I, Ferner M. Prevalence of pain 6 months after surgery: a prospective observational study. BMC Anesthesiol. 2016 Oct 10;16(1):91. doi: 10.1186/s12871-016-0261-7. PMID 27724844